CLINICAL TRIAL: NCT03156972
Title: Assessment of Rheumatic Heart Disease Patients With Chronic Severe Mitral Regurge by Speckle Tracking Echocardiography for Proper Timing of Surgical Operation.
Brief Title: Speckle Tracking for Timing of Surgical Operation in Severe Mitral Regurge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed mahmoud mohammed othman (Other)
Responsible Party: Sponsor-Investigator, Mohammed mahmoud mohammed othman, Assessment of rheumatic heart disease patients with chronic severe mitral regurge by Speckle Tracking Echocardiography for proper timing of surgical operation, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ossman231speckle
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group a (Active Comparator)
  Interventions: Procedure: Replacment of mitral valve
- Group b (Active Comparator)
  Interventions: Procedure: Replacment of mitral valve

INTERVENTIONS:
Procedure: Replacment of mitral valve — Mitral valve replacment by prothsis

SUMMARY:
Rhumatic heart disease patients with mitral regurge untile know had adibat for timming of surgical interferance our study aim to solve this problme using a new technic in echocardiography called speckle tracking which is more accurate in estimating a changes occure to myocyte of the heart and so chosing the proper time for surgery

ELIGIBILITY:
Inclusion Criteria:

* rhuematic heart disease with severe mitral regurge

Exclusion Criteria:

* non rheumatic mitral regurge

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Timing of surgical operation in patients with chronic severe mitral regurge | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aly, Prof, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No